CLINICAL TRIAL: NCT02480634
Title: Zoledronic Acid Combined Radiotherapy for Bone Metastasis of Non-small Cell Lung Cancer: A Non-inferiority, Randomized, Open, Parallel and Controlled Prospective Clinical Study
Brief Title: Zoledronic Acid Combined Radiotherapy for Bone Metastasis of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Wang Ge, Botanic physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPRA-1023-SK
Record Dates: First submitted 2015-03-17; First posted 2015-06-24 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Non-small Cell Lung Cancer; Bone Metastasis
Keywords: zoledronic acid; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Zoledronic Acid; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose group (Active Comparator): Zoledronic acid 4 mg + 0.9% sodium chloride injection 100 ml intravenous drip more than 15 min, 28 days for a transfusion cycle , a total of six cycle，Radiotherapy dose: 30Gy/10f
  Interventions: Drug: Zoledronic acid; Radiation: Radiotherapy
- Low dose group (Experimental): Zoledronic acid 4 mg + 0.9% sodium chloride injection 100 ml intravenous drip more than 15 min, 28 days for a transfusion cycle, a total of six cycle，Radiotherapy dose: 15Gy/5f
  Interventions: Drug: Zoledronic acid; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Zoledronic acid — Comparison the curative effect of the high does radiotherapy and low does therapy after use the Zoledronic acid
  Other Names: Zometa
Radiation: Radiotherapy — High dose：30Gy/10f Low dose：15Gy/5f

SUMMARY:
This study will give comparison of the bone pain remission and the adverse reaction of Zoledronic acid combine with High dose fractionation radiotherapy(30Gy/10f) and Zoledronic acid combine with low dose fractionation radiotherapy(15Gy/5f) . The purpose of this trial is to prove whether Zoledronic acid combine radiotherapy can reduce radiotherapy dose in treatment of non-small cell lung cancer bone metastasis'pain relief or not.

DETAILED DESCRIPTION:
Further study details as provided by oncology center of Daping hospital

ELIGIBILITY:
Inclusion Criteria:

* Pathology or cytology was diagnosed with non-small cell lung cancer, and bone metastases was confirmed by CT or MRI , and the patients have to need intervention treatment.
* VAS score>2 points.
* No paraplegia,
* No pathological fractures of bone related events which require surgical intervention,
* No major organ dysfunction,laboratory indexes meet the following requirements: Haemamoeba >4.0 x 10^9/L, Neutrophile granulocyte > 2 x 10^9/L, the platelet count>100 x 10^9/L, hemoglobin>100 g/L; Liver result: the serum bilirubin is lower than normal ceiling; ALT and AST is lower than the maximum normal 1.5 times; Cr<265 umol/l or 3.0 mg/dl, creatinine clearance>60 ml/min.

Exclusion Criteria:

* The patients who have allergy of Bisphosphonates and zoledronate.
* The patients who receive Molecular targeted therapy and chemotherapy within one month，The patients who receive Calcitonin and Aminoglycoside therapy in one week.
* The patients who receive Pamidronic Acid in 28 days，The patients original sites receive radiotherapy before.
* The patients who have history of thyroid surgery，receive tooth extraction in 2 weeks，and have been suffered from Bone Fracture and paraplegia.
* The patients who have Serious internal medicine diseases and acute infection.
* The patients With a history of psychiatric
* Pregnancy or breast-feeding women, men have fertility requirements
* Patients within clinical trials or not more than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants reach objective response | Up to 1 month
  Objective response is defined as the patients bone pain relief reach PR(Partial remission) or CR(Complete remission).and Objective response rate is defined as Objective response patients'percentage in total patients.
  Time evaluation points 1 month is the time after radiotherapy.

SECONDARY OUTCOMES:
Percentage of Participants occur bone pain recurrence at 1 to 12 month after radiotherapy. | every months up to the 12th month after treatment
  Bone pain Recurrence is defined as the time of the original parts again pain and the VAS is more than 4 points.
Pain relief time in/after treatment | everyday in treatment and every months up to 12 monthes
  Pain relief time is defined as the time of the VAS(Visual analogue scale) score reduce 2 points or the analgesic reduce 25% after the radiotherapy Time evaluation points :when patients in treatment ,we shall evaluate pain scores everyday ; when patients after treatment,we shall evluate pain scores every month.
Incidence of SRE(Skeletal-related events) again in Participants | every monthes up to the 12th month after treatment
  Incidence of SRE again is defined as the Participants occur SRE events after treatment.
  Time evaluation points :When patients were after treat,we shall evaluate whether occur SRE again every month.
Security of the therapy | everyday in treatment and every months up to the 12th month after treatment
  Time evaluation points :when patients were in treatment ,we shall evaluate the toxicity everyday ; when patients were after treatment,we shall evluate toxicity every month.
  Method：Using RTOG acute radiation injury grading assessment and RTOG / EORTC late radiation injury grading for radiotherapy toxicity，CTCAE V3.0 for Adverse drug reactions.
Percentage of the osteogenic and the osteolytic sites reach objective response | every months up to the 12th month
Kaplan-Meier Estimates for Overall Survival after bone metastases | every months up to the 12th month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ge Wang, Doctor, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University

REFERENCES:
- [Background] Akbar RA, Gosh SK, Khalil S, ul Haq SM. Zoledronic acid in metastatic bone disease: an audit based discussion. J Ayub Med Coll Abbottabad. 2010 Jul-Sep;22(3):5-7. PMID 22338405
- [Background] Wu JS, Wong R, Johnston M, Bezjak A, Whelan T; Cancer Care Ontario Practice Guidelines Initiative Supportive Care Group. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):594-605. doi: 10.1016/s0360-3016(02)04147-0. PMID 12573746
- [Background] Chow E, Wu JS, Hoskin P, Coia LR, Bentzen SM, Blitzer PH. International consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Radiother Oncol. 2002 Sep;64(3):275-80. doi: 10.1016/s0167-8140(02)00170-6. PMID 12242115
- [Background] Chow E, Hoskin P, Mitera G, Zeng L, Lutz S, Roos D, Hahn C, van der Linden Y, Hartsell W, Kumar E; International Bone Metastases Consensus Working Party. Update of the international consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12. PMID 21489705
- [Background] Dennis K, Makhani L, Zeng L, Lam H, Chow E. Single fraction conventional external beam radiation therapy for bone metastases: a systematic review of randomised controlled trials. Radiother Oncol. 2013 Jan;106(1):5-14. doi: 10.1016/j.radonc.2012.12.009. Epub 2013 Jan 13. PMID 23321492
- [Background] Luo KW, Ko CH, Yue GG, Lee MY, Siu WS, Lee JK, Shum WT, Fung KP, Leung PC, Li G, Evdokiou A, Lau CB. Anti-tumor and anti-osteolysis effects of the metronomic use of zoledronic acid in primary and metastatic breast cancer mouse models. Cancer Lett. 2013 Oct 1;339(1):42-8. doi: 10.1016/j.canlet.2013.07.024. Epub 2013 Jul 26. PMID 23896464
- [Background] Denham JW, Wilcox C, Joseph D, Spry NA, Lamb DS, Tai KH, Matthews J, Atkinson C, Turner S, Christie D, Gogna NK, Kenny L, Duchesne G, Delahunt B, McElduff P. Quality of life in men with locally advanced prostate cancer treated with leuprorelin and radiotherapy with or without zoledronic acid (TROG 03.04 RADAR): secondary endpoints from a randomised phase 3 factorial trial. Lancet Oncol. 2012 Dec;13(12):1260-70. doi: 10.1016/S1470-2045(12)70423-0. Epub 2012 Nov 12. PMID 23151431
- [Background] Denham JW, Joseph D, Lamb DS, Spry NA, Duchesne G, Matthews J, Atkinson C, Tai KH, Christie D, Kenny L, Turner S, Gogna NK, Diamond T, Delahunt B, Oldmeadow C, Attia J, Steigler A. Short-term androgen suppression and radiotherapy versus intermediate-term androgen suppression and radiotherapy, with or without zoledronic acid, in men with locally advanced prostate cancer (TROG 03.04 RADAR): an open-label, randomised, phase 3 factorial trial. Lancet Oncol. 2014 Sep;15(10):1076-89. doi: 10.1016/S1470-2045(14)70328-6. Epub 2014 Aug 14. PMID 25130995
- [Background] Deberne M, Ropert S, Billemont B, Daniel C, Chapron J, Goldwasser F. Inaugural bone metastases in non-small cell lung cancer: a specific prognostic entity? BMC Cancer. 2014 Jun 10;14:416. doi: 10.1186/1471-2407-14-416. PMID 24913188
- [Background] Peng H, Ma M, Han B. [Survival analysis of 1,742 patients with stage IV non-small cell lung cancer]. Zhongguo Fei Ai Za Zhi. 2011 Apr;14(4):362-6. doi: 10.3779/j.issn.1009-3419.2011.04.11. Chinese. PMID 21496437
- [Background] Bae HM, Lee SH, Kim TM, Kim DW, Yang SC, Wu HG, Kim YW, Heo DS. Prognostic factors for non-small cell lung cancer with bone metastasis at the time of diagnosis. Lung Cancer. 2012 Sep;77(3):572-7. doi: 10.1016/j.lungcan.2012.05.094. Epub 2012 Jun 4. PMID 22672969
- [Background] Nakamura N, Shikama N, Wada H, Harada H, Nozaki M, Nagakura H, Tago M, Oguchi M, Uchida N; Japanese Radiation Oncology Study Group Working Subgroup of Palliative Radiotherapy. Patterns of practice in palliative radiotherapy for painful bone metastases: a survey in Japan. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):e117-20. doi: 10.1016/j.ijrobp.2011.11.075. Epub 2012 Feb 28. PMID 22381902
- [Background] Brown JE, Cook RJ, Major P, Lipton A, Saad F, Smith M, Lee KA, Zheng M, Hei YJ, Coleman RE. Bone turnover markers as predictors of skeletal complications in prostate cancer, lung cancer, and other solid tumors. J Natl Cancer Inst. 2005 Jan 5;97(1):59-69. doi: 10.1093/jnci/dji002. PMID 15632381
- [Background] Sun JM, Ahn JS, Lee S, Kim JA, Lee J, Park YH, Park HC, Ahn MJ, Ahn YC, Park K. Predictors of skeletal-related events in non-small cell lung cancer patients with bone metastases. Lung Cancer. 2011 Jan;71(1):89-93. doi: 10.1016/j.lungcan.2010.04.003. Epub 2010 Jul 3. PMID 20598769
- [Background] Zhang L, Hou X, Lu S, Rao H, Hou J, Luo R, Huang H, Zhao H, Jian H, Chen Z, Liao M, Wang X. Predictive significance of bone sialoprotein and osteopontin for bone metastases in resected Chinese non-small-cell lung cancer patients: a large cohort retrospective study. Lung Cancer. 2010 Jan;67(1):114-9. doi: 10.1016/j.lungcan.2009.03.017. PMID 19376608
- [Background] Dennis K, Wong K, Zhang L, Culleton S, Nguyen J, Holden L, Jon F, Tsao M, Danjoux C, Barnes E, Sahgal A, Zeng L, Koo K, Chow E. Palliative radiotherapy for bone metastases in the last 3 months of life: worthwhile or futile? Clin Oncol (R Coll Radiol). 2011 Dec;23(10):709-15. doi: 10.1016/j.clon.2011.05.004. Epub 2011 Jun 12. PMID 21665446
- [Background] Hirsh V. Skeletal disease contributes substantially to morbidity and mortality in patients with lung cancer. Clin Lung Cancer. 2009 Jul;10(4):223-9. doi: 10.3816/CLC.2009.n.030. PMID 19632938
- [Background] Pandya KJ, Gajra A, Warsi GM, Argonza-Aviles E, Ericson SG, Wozniak AJ. Multicenter, randomized, phase 2 study of zoledronic acid in combination with docetaxel and carboplatin in patients with unresectable stage IIIB or stage IV non-small cell lung cancer. Lung Cancer. 2010 Mar;67(3):330-8. doi: 10.1016/j.lungcan.2009.04.020. Epub 2009 Jun 2. PMID 19493585
- [Background] Cheon PM, Pulenzas N, Zhang L, Mauti E, Wong E, Thavarajah N, Tsao M, Danjoux C, Holden L, DeAngelis C, Chow E. Fatigue scores in patients receiving palliative radiotherapy for painful bone metastases. Support Care Cancer. 2015 Jul;23(7):2097-103. doi: 10.1007/s00520-014-2561-0. Epub 2014 Dec 24. PMID 25533579
- [Background] Cole DJ. A randomized trial of a single treatment versus conventional fractionation in the palliative radiotherapy of painful bone metastases. Clin Oncol (R Coll Radiol). 1989 Nov;1(2):59-62. doi: 10.1016/s0936-6555(89)80035-4. PMID 2484789
- [Background] Wu JS, Bezjak A, Chow E, Kirkbride P. Primary treatment endpoint following palliative radiotherapy for painful bone metastases: need for a consensus definition? Clin Oncol (R Coll Radiol). 2002 Feb;14(1):70-7. doi: 10.1053/clon.2001.0012. PMID 11899906
- [Background] Popovic M, den Hartogh M, Zhang L, Poon M, Lam H, Bedard G, Pulenzas N, Lechner B, Chow E. Review of international patterns of practice for the treatment of painful bone metastases with palliative radiotherapy from 1993 to 2013. Radiother Oncol. 2014 Apr;111(1):11-7. doi: 10.1016/j.radonc.2014.01.015. Epub 2014 Feb 20. PMID 24560750
- [Background] Westhoff PG, de Graeff A, Reyners AK, Monninkhof EM, Rodenhuis CC, van Vulpen M, Leer JW, Marijnen CA, van der Linden YM; Dutch Bone Metastasis Study Group. Effect of age on response to palliative radiotherapy and quality of life in patients with painful bone metastases. Radiother Oncol. 2014 May;111(2):264-9. doi: 10.1016/j.radonc.2014.03.017. Epub 2014 Apr 17. PMID 24746581
- [Background] Konski A, James J, Hartsell W, Leibenhaut MH, Janjan N, Curran W, Roach M, Watkins-Bruner D. Economic analysis of radiation therapy oncology group 97-14: multiple versus single fraction radiation treatment of patients with bone metastases. Am J Clin Oncol. 2009 Aug;32(4):423-8. doi: 10.1097/COC.0b013e31818da9f7. PMID 19546803
- [Background] Li YY, Chang JW, Chou WC, Liaw CC, Wang HM, Huang JS, Wang CH, Yeh KY. Zoledronic acid is unable to induce apoptosis, but slows tumor growth and prolongs survival for non-small-cell lung cancers. Lung Cancer. 2008 Feb;59(2):180-91. doi: 10.1016/j.lungcan.2007.08.026. Epub 2007 Sep 27. PMID 17900752
- [Background] Lipton A. Treatment of bone metastases and bone pain with bisphosphonates. Support Cancer Ther. 2007 Jan 1;4(2):92-100. doi: 10.3816/SCT.2007.n.003. PMID 18632473
- [Background] Henk H, Teitelbaum A, Kaura S. Evaluation of the clinical benefit of long-term (beyond 2 years) treatment of skeletal-related events in advanced cancers with zoledronic acid. Curr Med Res Opin. 2012 Jul;28(7):1119-27. doi: 10.1185/03007995.2012.689254. Epub 2012 May 17. PMID 22536885
- [Background] Wang Z, Qiao D, Lu Y, Curtis D, Wen X, Yao Y, Zhao H. Systematic literature review and network meta-analysis comparing bone-targeted agents for the prevention of skeletal-related events in cancer patients with bone metastasis. Oncologist. 2015 Apr;20(4):440-9. doi: 10.1634/theoncologist.2014-0328. Epub 2015 Mar 2. PMID 25732263
- [Background] Saad F, Chen YM, Gleason DM, Chin J. Continuing benefit of zoledronic acid in preventing skeletal complications in patients with bone metastases. Clin Genitourin Cancer. 2007 Sep;5(6):390-6. doi: 10.3816/CGC.2007.n.022. PMID 17956712
- [Result] Takeda N, Isu K, Hiraga H, Shinohara N, Minami A, Kamata H. Zoledronic acid enhances the effect of radiotherapy for bone metastases from renal cell carcinomas: more than a 24-month median follow-up. J Orthop Sci. 2012 Nov;17(6):770-4. doi: 10.1007/s00776-012-0294-9. Epub 2012 Oct 2. PMID 23053582
- [Result] Atahan L, Yildiz F, Cengiz M, Kaplan B, Ozkan M, Yazici G, Gundog M, Haydaroglu A, Korcum AF, Sengoz M, Dincer M, Akmansu M, Engin K, Hayran M. Zoledronic acid concurrent with either high- or reduced-dose palliative radiotherapy in the management of the breast cancer patients with bone metastases: a phase IV randomized clinical study. Support Care Cancer. 2010 Jun;18(6):691-8. doi: 10.1007/s00520-009-0663-x. Epub 2009 May 31. PMID 19484483